CLINICAL TRIAL: NCT03381950
Title: Chronic Kidney Disease - Renal Epidemiology and Information Network: The CKD-REIN Cohort
Brief Title: Chronic Kidney Disease - Renal Epidemiology and Information Network
Acronym: CKD-REIN
Status: Active, not recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Université Paris-Sud (Other); Agence de La Biomédecine (Other Government); Arbor Research Collaborative for Health (Other); Hospital Ambroise Paré Paris (Other); Centre Hospitalier Lyon Sud (Other); Central Hospital, Nancy, France (Other); Institut de Formation et de Recherche sur les Organisations Sanitaires et Sociales (Unknown); Biobanque de Picardie (Unknown); Centre National de Génotypage (Other); Institut des Maladies Métaboliques et Cardiovasculaires (Unknown); Etablissement Français du Sang (Other); Amiens University Hospital (Other); University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: C12-30
Record Dates: First submitted 2017-12-11; First posted 2017-12-22 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Renal Insufficiency, Chronic
Keywords: chronic kidney disease; prospective cohort study; risk profile; patient-reported-outcomes
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma and urine samples are collected and stored on all patients at enrollment and study end, and in a subsample of 1,200 at 2-year follow-up.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preserving kidney function and improving the transition from CKD to End stage renal disease (ESRD) is a research and healthcare challenge. The Chronic Kidney Disease-Renal Epidemiology and Information Network (CKD-REIN) cohort was established to identify the determinants, biomarkers and practice patterns associated with chronic kidney disease outcomes. The study includes 3,033 adult patients with moderate to advanced CKD from a representative sample of 40 nephrology clinics in France with respect to regions and legal status. Patients are recruited during a routine visit and followed up for 5 years, before and after starting renal replacement therapy. Patient-level clinical, biological, and lifestyle data are collected annually, as well as provider-level data on clinical practices, coordinated with the International Chronic Kidney Disease Outcomes and Practice Pattern Study (CKDopps). Blood and urine samples are stored in a biobank. The overall objective is to develop a research platform to address key questions regarding the determinants and biomarkers associated with adverse outcomes in CKD and to assess its effective management. It has the following hypotheses and specific aims:

1. to evaluate a large set of social, environmental, bioclinical, and genetic factors, and their interactions in relation with CKD outcomes including progression to ESRD, mortality, metabolic and vascular complications, and the onset of a number of chronic and acute events;
2. to assess several new biomarkers to predict adverse outcomes of CKD and its complications;
3. to evaluate the associations of provider practices (management of hypertension, anemia, nutritional abnormalities, mineral and bone disorder, nutritional status, timing of dialysis initiation and transplant wait-listing) with achievement of clinical practice guidelines, clinical and patient-reported outcomes (PRO).
4. to evaluate the associations of health care organization and clinic services (e.g., for nutrition, educational programs) with clinical and patient-reported outcomes, and achievement of clinical practice guidelines;
5. to estimate the relative cost-effectiveness of different provider practices and clinic services.

DETAILED DESCRIPTION:
All cohort participants are assessed annually for at least 5 years, until 6 months after the start of renal replacement therapy.

Each year, data are collected from both medical records and patients interview and self-administrated questionnaires are asked to report clinical events.

Interviews and routine biological measurements are repeated annually.

CKD-REIN is funded by the Agence Nationale de la Recherche through the 2010 'Cohortes-Investissements d'Avenir' programme and by the 2010 national Programme Hospitalier de Recherche Clinique.

CKD-REIN is also supported through a public-private partnership with Amgen, Fresenius Medical Care, and GlaxoSmithKline since 2012; Baxter and MerckSharp&Dohme-Chibret (France) from 2012 to 2017; LillyFrance since 2013; Otsuka Pharmaceutical since 2015; Vifor Fresenius since 2017; AstraZeneca since 2018; and Sanofi-Genzyme from 2012 to 2015.

ELIGIBILITY:
Inclusion Criteria:

* eGFR < 60 ml/min/1.73m2 for at least 1 month
* no prior chronic dialysis or transplantation
* Written Signed consent form

Exclusion Criteria:

* Age <18 yrs old,
* Pregnant female,
* patients who plan to move
* Unable to give inform consent,
* Decline to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CKD Stage 3-5 (eGFR <60 ml/min/1.73m2, not on dialysis or with kidney transplant) receiving nephrology care
Sampling Method: Non-Probability Sample
Enrollment: 3033 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of end-stage renal disease (ESRD) | up to 5 years
  Dialysis, transplantation, conservative care management

SECONDARY OUTCOMES:
Mortality | up to 5 years
  Specific and all-cause mortality
Incidence of major CKD events including acute kidney injury, cardiovascular and metabolic complications | up to 5 years
Incidence of major adverse events including infections, cancer, mineral and bone disease, anemia, nutitional status, hospitalizations | up to 5 years
Prescription drug use | up to 5 years
  For each drug prescription, the trade name, international non-proprietary name, ATC class, unit dose, defined daily dose, pharmaceutical formulation, and administration route are recorded. A linkage with the drug reimbursement files from the health insurance will be also performed.
Health-related Quality of life | up to 5 years
  Assessed by the Kidney Disease Quality of Life (KDQOL™) scale. It is a measure of kidney disease-related quality of life that comprises four subscales: Generic core [Physical Component Summary (PCS) and Mental Component Summary (MCS)]; Symptoms/Problems; Burden of Kidney Disease, and Effects of Kidney Disease. Scores of each subscale are calculated, ranged from 0 to 100, with higher scores reflecting better quality of life.
Depression | up to 5 years
  Assessed by the 10-item Center for Epidemiologic Studies Depression Scale (CESD). It is a screening test for depression and depressive disorder. A total score is reported.The possible range is 0 to 30, with the higher scores indicating more depression symptoms.
Cognitive function | up to 5 years
  The 30-item minimental status examination (MMSE) is a practical tool for evaluating cognitive status. A total score is reported, ranged from 0 to 30, with the higher scores indicating less cognitive impairment.
Physical Activity | up to 5 years
  The French translation of the Global Physical Activity Questionnaire (Version 2.0) is used to gather information on the time spent in moderate and vigorous physical activity and in sedentary behavior. The GPAQ contains 16 items designed to assess the frequency and duration of physical activity in 3 domains: during work, transportation, and leisure time as well as time spent sitting during a typical week. It distinguishes physical activity duration by min/day and min/week for each physical activity domain, which allows for calculating the energy expenditure scored in metabolic equivalent tasks (METs). According to duration and energy expenditure, physical activity level was classified as low, moderate, and high.
Family relationships | up to 5 years
  Assessed by the Family Relationships Index (FRI). the FRI provides a brief measure of family relations by assessing the way people currently perceive and describe their family. The scale consists of 12 items. Each item is coded from 1 to 4. A validation study of this questionnaire is planned.
Sleep disorders | up to 5 years
Women's health | up to 5 years
  Set of questions regarding the menopause, menstrual cycle and contraception, and past/in progress pregnancies.
Cost effectiveness of different treatment practices and services | up to 5 years
  Several data sources will be used to estimate the cost of different treatment practices and services.
  Patient-Level: key resource utilization indicators (e.g., hospitalization, clinic visits, prescription drug use), and procedures for costing these measures.
  Clinic-level: The net costs of different treatment practices as well as structural characteristics (such as number of beds of the hospital, number of wards, number of hierarchical levels, for-profit or non for-profit status, teaching or not teaching hospital, spatial organization).

CONTACTS AND LOCATIONS:
Overall Officials: Bénédicte Stengel, MD, Principal Investigator — Inserm U1018, UPS-UVSQ, CESP, Renal and Cardiovascular Epidemiology team, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stengel B, Combe C, Jacquelinet C, Briancon S, Fouque D, Laville M, Frimat L, Pascal C, Herpe YE, Deleuze JF, Schanstra J, Pisoni RL, Robinson BM, Massy ZA. The French Chronic Kidney Disease-Renal Epidemiology and Information Network (CKD-REIN) cohort study. Nephrol Dial Transplant. 2014 Aug;29(8):1500-7. doi: 10.1093/ndt/gft388. Epub 2013 Sep 24. PMID 24064325
- [Background] Stengel B, Combe C, Jacquelinet C, Briancon S, Fouque D, Laville M, Frimat L, Pascal C, Herpe YE, Morel P, Deleuze JF, Schanstra JP, Pisoni RL, Robinson BM, Massy ZA. [The French Chronic Kidney Disease-Renal Epidemiology and Information Network (CKD-REIN) cohort study: To better understand chronic kidney disease]. Nephrol Ther. 2016 Apr;12 Suppl 1:S49-56. doi: 10.1016/j.nephro.2016.01.005. Epub 2016 Mar 11. French. PMID 26976057
- [Background] Laville SM, Stengel B, Massy ZA, Liabeuf S. Reply to "Restricting maintenance allopurinol dose according to kidney function in patients with gout is inappropriate!" by Stamp et al. Br J Clin Pharmacol. 2019 Jun;85(6):1380-1381. doi: 10.1111/bcp.13924. Epub 2019 Apr 13. No abstract available. PMID 30980562
- [Result] Affret A, Wagner S, El Fatouhi D, Dow C, Correia E, Niravong M, Clavel-Chapelon F, De Chefdebien J, Fouque D, Stengel B; CKD-REIN study investigators; Boutron-Ruault MC, Fagherazzi G. Validity and reproducibility of a short food frequency questionnaire among patients with chronic kidney disease. BMC Nephrol. 2017 Sep 15;18(1):297. doi: 10.1186/s12882-017-0695-2. PMID 28915857
- [Result] Villain C, Metzger M, Combe C, Fouque D, Frimat L, Jacquelinet C, Laville M, Briancon S, Klein J, Schanstra JP, Robinson BM, Mansencal N, Stengel B, Massy ZA. Prevalence of atheromatous and non-atheromatous cardiovascular disease by age in chronic kidney disease. Nephrol Dial Transplant. 2020 May 1;35(5):827-836. doi: 10.1093/ndt/gfy277. PMID 30169874
- [Result] Laville SM, Metzger M, Stengel B, Jacquelinet C, Combe C, Fouque D, Laville M, Frimat L, Ayav C, Speyer E, Robinson BM, Massy ZA, Liabeuf S; Chronic Kidney Disease-Renal Epidemiology and Information Network (CKD-REIN) Study Collaborators. Evaluation of the adequacy of drug prescriptions in patients with chronic kidney disease: results from the CKD-REIN cohort. Br J Clin Pharmacol. 2018 Dec;84(12):2811-2823. doi: 10.1111/bcp.13738. Epub 2018 Sep 24. PMID 30110711
- [Result] Balkau B, Metzger M, Andreelli F, Frimat L, Speyer E, Combe C, Laville M, Jacquelinet C, Briancon S, Ayav C, Massy Z, Pisoni RL, Stengel B, Fouque D. Impact of sex and glucose-lowering treatments on hypoglycaemic symptoms in people with type 2 diabetes and chronic kidney disease. The French Chronic Kidney Disease - Renal Epidemiology and Information Network (CKD-REIN) Study. Diabetes Metab. 2019 Apr;45(2):175-183. doi: 10.1016/j.diabet.2018.03.007. Epub 2018 Apr 6. PMID 29706470
- [Result] Stengel B, Metzger M, Combe C, Jacquelinet C, Briancon S, Ayav C, Fouque D, Laville M, Frimat L, Pascal C, Herpe YE, Morel P, Deleuze JF, Schanstra JP, Lange C, Legrand K, Speyer E, Liabeuf S, Robinson BM, Massy ZA. Risk profile, quality of life and care of patients with moderate and advanced CKD: The French CKD-REIN Cohort Study. Nephrol Dial Transplant. 2019 Feb 1;34(2):277-286. doi: 10.1093/ndt/gfy058. PMID 29635335
- [Result] Schweitzer ML, Stengel B, Legrand K, Briancon S, Jacquelinet C, Combe C, Fouque D, Massy ZA, Laville M, Frimat L, Ayav C. Obesity phenotype and patient-reported outcomes in moderate and severe chronic kidney disease: a cross-sectional study from the CKD-REIN cohort study. Qual Life Res. 2019 Jul;28(7):1873-1883. doi: 10.1007/s11136-019-02110-2. Epub 2019 Jan 18. PMID 30659448
- [Result] Sukul N, Speyer E, Tu C, Bieber BA, Li Y, Lopes AA, Asahi K, Mariani L, Laville M, Rayner HC, Stengel B, Robinson BM, Pisoni RL; CKDopps and CKD-REIN investigators. Pruritus and Patient Reported Outcomes in Non-Dialysis CKD. Clin J Am Soc Nephrol. 2019 May 7;14(5):673-681. doi: 10.2215/CJN.09600818. Epub 2019 Apr 11. PMID 30975656
- [Result] Liabeuf S, McCullough K, Young EW, Pisoni R, Zee J, Reichel H, Pecoits-Filho R, Port FK, Stengel B, Csomor PA, Metzger M, Robinson B, Massy ZA. International variation in the management of mineral bone disorder in patients with chronic kidney disease: Results from CKDopps. Bone. 2019 Dec;129:115058. doi: 10.1016/j.bone.2019.115058. Epub 2019 Sep 4. PMID 31493530
- [Result] Pecoits-Filho R, Fliser D, Tu C, Zee J, Bieber B, Wong MMY, Port F, Combe C, Lopes AA, Reichel H, Narita I, Stengel B, Robinson BM, Massy Z; CKDopps Investigators. Prescription of renin-angiotensin-aldosterone system inhibitors (RAASi) and its determinants in patients with advanced CKD under nephrologist care. J Clin Hypertens (Greenwich). 2019 Jul;21(7):991-1001. doi: 10.1111/jch.13563. Epub 2019 Jun 6. PMID 31169352
- [Derived] Laville SM, Jaisson S, Gillery P, Okwieka A, Alencar de Pinho N, Combe C, Mansencal N, Massy ZA, Liabeuf S; CKD-REIN study collaborators. Homocitrulline Is Associated with Cardiovascular Outcomes in Nondialysis Patients with CKD. Kidney360. 2025 Apr 1;6(8):1328-1337. doi: 10.34067/KID.0000000797. PMID 40168087
- [Derived] El Chamieh C, Larabi IA, Laville SM, Jacquelinet C, Combe C, Fouque D, Laville M, Frimat L, Pecoits-Filho R, Lange C, Stengel B, Alencar De Pinho N, Alvarez JC, Massy ZA, Liabeuf S; Chronic Kidney Disease-Renal Epidemiology and Information Network (CKD-REIN) Study Group. Proton-Pump Inhibitors and Serum Concentrations of Uremic Toxins in Patients with Chronic Kidney Disease. Toxins (Basel). 2023 Apr 7;15(4):276. doi: 10.3390/toxins15040276. PMID 37104214
- [Derived] Montalescot L, Dorard G, Speyer E, Legrand K, Ayav C, Combe C, Stengel B, Untas A. The experience of relatives and friends of patients with moderate to advanced chronic kidney disease: Insights from the CKD-REIN cohort study. Br J Health Psychol. 2023 Nov;28(4):930-951. doi: 10.1111/bjhp.12662. Epub 2023 Apr 20. PMID 37080946
- [Derived] Pepin M, Levassort H, Boucquemont J, Lambert O, Alencar de Pinho N, Turinici M, Helmer C, Metzger M, Cheddani L, Frimat L, Combe C, Fouque D, Laville M, Ayav C, Liabeuf S, Jacquelinet C, Teillet L, Stengel B, Massy ZA; CKD-REIN Study Collaborators. Cognitive performance is associated with glomerular filtration rate in patients with chronic kidney disease: results from the CKD-REIN cohort. J Neurol Neurosurg Psychiatry. 2023 Jun;94(6):457-466. doi: 10.1136/jnnp-2022-330347. Epub 2023 Jan 24. PMID 36693722
- [Derived] Wagner S, Merkling T, Metzger M, Koppe L, Laville M, Boutron-Ruault MC, Frimat L, Combe C, Massy ZA, Stengel B, Fouque D. Probiotic Intake and Inflammation in Patients With Chronic Kidney Disease: An Analysis of the CKD-REIN Cohort. Front Nutr. 2022 Mar 30;9:772596. doi: 10.3389/fnut.2022.772596. eCollection 2022. PMID 35433774
- [Derived] Montalescot L, Speyer E, Legrand K, Ayav C, Combe C, Stengel B, Untas A. Reliability and validity of the French adaptation of the Family Relationship Index-short form in patients' with chronic kidney disease. J Health Psychol. 2022 Jan;27(1):166-175. doi: 10.1177/1359105320949921. Epub 2020 Aug 10. PMID 32772863
- [Derived] Laville SM, Gras-Champel V, Moragny J, Metzger M, Jacquelinet C, Combe C, Fouque D, Laville M, Frimat L, Robinson BM, Stengel B, Massy ZA, Liabeuf S; Chronic Kidney Disease-Renal Epidemiology and Information Network (CKD-REIN) Study Group. Adverse Drug Reactions in Patients with CKD. Clin J Am Soc Nephrol. 2020 Aug 7;15(8):1090-1102. doi: 10.2215/CJN.01030120. Epub 2020 Jul 1. PMID 32611662
- See also: The CKD-REIN Website — https://ckdrein.inserm.fr